CLINICAL TRIAL: NCT01308645
Title: PhaseⅡ, Open Label, Clinical Trial to Investigate Safety and Efficacy of SB Injection in Patients With Advanced or Primary Hepatocellular Carcinoma
Brief Title: Evaluating the Safety and Efficacy of SB Injection in Patients With Advanced or Primary Hepatocellular Carcinoma (HCC)
Acronym: HCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: SBPharmaceutical IND, Co., LTD (Industry)
Responsible Party: Lee Dong-heum / executive director, SBPharmaceutical IND, Co., LTD
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SB Injection HCC
Record Dates: First submitted 2011-03-02; First posted 2011-03-04 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: SBP Injection; HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: SB injection — Infusion SB injection of 21.87 ml/m^2, IV route, 24 times for 4 months

SUMMARY:
The purpose of this study is to determine efficacy of SB injection in Hepatocellular Carcinoma (HCC).

DETAILED DESCRIPTION:
All eligible patients will receive SB injection therapy for 6 cycles (14~21 days for each cycle). Efficacy wll be evaluated every 3 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 years or over
2. Patients with Hepatocellular carcinoma progression (HCC) and primary liver cancer as a diagnostic imaging test (eg, X-ray, CT, scan, ultrasound) can be measured in patients with a lesion
3. Directly to standard therapy (surgery, RF ablation, TACE) is not possible, patients with advanced liver cancer. However, the standard treatment of the subject or subjects entirely voluntary participation of subjects participating at the discretion of the doctor or researcher can be deemed included in the selected target.
4. Life expectancy ≥ 5 months
5. ECOG status 0, 1, 2 patients
6. Child-Pugh classification A, B patients
7. PLT 70,000, ANC 1,000 or more patients (OT / PT <upper normal limit x 5.0, Bilirubin <upper normal limit x 3.0)
8. Female volunteers admitted to the study must be using a reliable means of contraception and must have a negative blood or urine pregnancy test at least 7 days ago
9. Patients or their legal representatives who have signed the informed consent form

Exclusion Criteria:

1. Last 4 weeks the patients who had participated in another clinical trial
2. Last 4 weeks the patients who received chemotherapy
3. Associated with hepatocellular carcinoma in patients with a history of malignant tumor
4. Hepatectomy or liver transplantation patients who received treatment.
5. Active systemic infection requiring medical treatment
6. Uncontrolled hypertension or diabetes mellitus.
7. Clinically Significant cardiac disease (myocardial infarction / angina / severe arrhythmia / congestive heart failure)
8. Autoimmune diseases (systemic lupus erythematosus: SLE / rheumatoid arthritis / myasthenia gravis) and the patients currently being treated
9. Presence or history of malignancy other than Hepatocellular carcinoma within 5 years
10. Patients who have history of allergy with this investigational drug.
11. Obvious cognitive or physical impairment that would prevent participation
12. Pregnancy, lactation period and don't using contraception earnest Patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-12 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Evaluating Tumor Response Rate | 4 Months

SECONDARY OUTCOMES:
Pain Scores on the Visual Analog Scale | 4 Months
Number of Participants with Adverse Events as a Measure of Safety and Tolerability scale | 4 Months
Determine duration of response rate by measuring time to progression | 4 Months

CONTACTS AND LOCATIONS:
Overall Officials: Lee Jin woo, Prof., Principal Investigator — Inha University Hospital
Locations (1):
- Inha University Hospital, Incheon, Jung-gu, South Korea

REFERENCES:
- See also: Link Text : SBP — http://www.sbp.com